CLINICAL TRIAL: NCT03361553
Title: Developing a Novel Clinical Tool to Evaluate Obstructive Sleep Apnea (OSA) with Airway Ultrasound
Brief Title: Obstructive Sleep Apnea Airway Evaluation
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 16-6160
Record Dates: First submitted 2017-11-14; First posted 2017-12-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Current practice guidelines recommend obstructive sleep apnea (OSA) patients to stay in the post anesthetic care unit (PACU) until the risk of respiratory depression has subsided. Inevitably, a greater demand on hospital resource utilization in these patients will increase health care cost. Polysomnography (PSG) and screening questionnaires can identify OSA but they are limited by accessibility and false positive results, respectively. Inaccurate OSA identification misguides postoperative surveillance plan. In contrast with MRI and CT scans, ultrasound is more accessible and more likely a practical tool for OSA screening. However, before clinical application, airway ultrasound (US) exam must undergo vigorous testing to check its utility, accuracy, inter-observer reliability and its ability to identify OSA and its severity.

DETAILED DESCRIPTION:
The investigators plan to recruit surgical patients at risk of OSA, exposed to sedatives,and/or general anesthesia. Surface ultrasound measurements will be conducted in a separate setting, and be correlated with the sleep study results, and a set of ultrasound parameters will be validated in this setting. Relevant clinical outcomes will be captured as well.

ELIGIBILITY:
Inclusion criteria

* age≥18
* ASA physical status I - IV;
* Suspected to have OSA for clinical reasons such as high risk on screening questionnaire i.e., a STOP-Bang score >3, and referred to have a sleep study for OSA diagnosis by the clinical team at any point of care during the perioperative period (such as the clinic using the screening tool, during or after surgery in the ward experiencing recurrent upper airway obstructive events, need for CPAP in the postoperative period and / or suspected to have obstructive airway events). Or;
* Patients who were recently diagnosed to have OSA and underwent a laboratory sleep study within the last year.
* Patients who were recently diagnosed to have OSA but are non-compliant with treatment. Compliance defined as: median nightly CPAP or APAP use > 70% of the nights, and for longer than 4 hours of nightly use during the last 3 months),43 or using oral appliance use (use > 70% of nights, and for longer than 4 hours of nightly use in the last 3 months.

Exclusion criteria

* failure to understand and provide consent
* past history of oral, head and neck surgery (e.g., OSA corrective surgery)
* active head & neck disease (e.g., cancer, infection and radiotherapy);
* inability to perform breathing tests per instruction
* Patients currently on treatment for OSA (as this may interfere with the upper airway dimensions and the US assessment may not be accurate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected / Recently diagnosed untreated Obstructive Sleep Apnea (amendment authorized 20/12/2017) / Non-compliant to OSA treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation of airway parameter measurements with Apnea-Hypopnea Index (AHI) values on Polysomnography (PSG) | 2 years
  The primary study outcome will be the discriminatory performance of each one of the airway parameters, against the OSA status (moderate/severe) as diagnosed by PSG.

SECONDARY OUTCOMES:
Feasibility of airway Ultrasound (US) examination; | 2 years
  1. The feasibility and efficiency of completing the US exam and reading the measurements;
  2. The inter-rater reliability for measuring each one of the airway parameters;
  3. The statistical association between each airway parameter and OSA severity level (none/mild/moderate/severe);
  4. The diagnostic accuracy for STOPBang (SB) score (ROC curve, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio, negative likelihood ratios, and diagnostic odds ratio (DOR) for different cut off levels);
  5. The correlation between each one of the airway parameters and the SB score; and
  6. The benefit of considering airway parameters in addition to SB in a prediction model for OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, Principal Investigator — Department of Anesthesia, Toronto Western Hospital- UHN, University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada